CLINICAL TRIAL: NCT05558007
Title: Phase 2 Clinical Trial to Evaluate Safety and Efficacy of BZ371A in a Gel Applied in Patients That Performed Radical Prostatectomy
Brief Title: Safety and Efficacy Evaluation of BZ371A Topically Applied on Prostatectomized Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biozeus Biopharmaceutical S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BZ371CLI004
Record Dates: First submitted 2022-09-22; First posted 2022-09-28 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy; Erectile Dysfunction; Prostate Cancer; Radical Prostatectomy
Keywords: Erectile Dysfunction; Radical Prostatectomy; Prostate Cancer
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Daily oral Tadalafil 5mg + Topical Placebo (Active Comparator): Patient that underwent Radical Prostatectomy will receive daily oral Tadalafil 5mg and topical placebo
  Interventions: Drug: Tadalafil 5mg; Drug: Topical Placebo
- Daily oral placebo + topical BZ371A (Experimental): Patient that underwent Radical Prostatectomy will receive daily oral placebo and topical BZ371A
  Interventions: Drug: BZ371A; Drug: Oral Placebo
- Daily oral Tadalafil 5mg + topical BZ371A (Active Comparator): Patient that underwent Radical Prostatectomy will receive daily oral Tadalafil 5mg and topical BZ371A
  Interventions: Drug: Tadalafil 5mg; Drug: BZ371A

INTERVENTIONS:
Drug: Tadalafil 5mg — Daily oral administration of tadalafil 5mg
  Other Names: Tadalafil
  Arms: Daily oral Tadalafil 5mg + Topical Placebo; Daily oral Tadalafil 5mg + topical BZ371A
Drug: BZ371A — Topical application of 1.5 mL of BZ371A in a concentration of 5mg/mL
  Arms: Daily oral Tadalafil 5mg + topical BZ371A; Daily oral placebo + topical BZ371A
Drug: Oral Placebo — Oral administration of a placebo pill
  Arms: Daily oral placebo + topical BZ371A
Drug: Topical Placebo — Topical application of 1.5 mL of placebo
  Arms: Daily oral Tadalafil 5mg + Topical Placebo

SUMMARY:
To determine efficacy, safety and tolerabiltiy of topically applied BZ371A in patients that experienced RP, in combination with daily tadalafil compared to placebo.

DETAILED DESCRIPTION:
Prostate cancer remains one of the most prevalent cancer in men. For its treatment, recent technological advances demonstrate that the most effective treatment is the Radical Prostatectomy (RP) procedure. However, although curative for Prostate Cancer, can result in damage to the cavernosal nerves.

The cavernosal autonomic nerves travel posterolaterally to the prostate to enter the penis and regulate blood flow and hence erection. Thus, damage caused by RP will affect NO tissue release and blood flow regulation, causing erectile dysfunction.

BZ371A has the ability to restore local blood flow regulation by a new and innovative mechanism of action and, therefore, has potential to be a supportive therapy for RP patients (restoring the erectile function).

Thus, this study aims to evaluate efficacy, safety and tolerabilty of BZ371A on the recovery of erectile function of patients that were underwent Radical Prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Men between the ages of 40 and 65 years;
2. Exclusive heterosexual men, regardless of race or social class.
3. RP due to prostate cancer without metastasis;
4. RP performed less than 60 days before the screening visit;
5. Erectile function prior to normal RP, defined as IIEF questionnaire with more than 22 points in domain A;
6. Stable sexual partner (more than 2 months prior to RP), and intention to maintain the relationship during the study.
7. Continuous use of 5mg Tadalafil from the 30th up to the 60th day after RP.

Exclusion Criteria:

1. Prostate cancer in TNM stage classified as T3 or T4.
2. Perineal and/or open RP;
3. Necessity of other therapy for prostate cancer than RP, including radiation therapy or hormone therapy;
4. Uncontrolled diabetes at screening visit (HbA1C > 10%);
5. Prior spinal cord injury with lower limb paralysis;
6. Current male hormone use, or hypogonadism, defined by total testosterone below 8 nmol/L (2300 pg/mL) or total testosterone between 8 and 11 nmol/L (2300 and 3170 pg/mL) and free testosterone < 220 pmol/L (< 64 ng/dL);
7. Patients with current depression, characterized by use or need for use of antidepressants.
8. Presence of genital lesions (such as severe penile fibrosis or Peyronie's disease) or active sexually transmitted disease (STD) (such as herpes, gonorrhea, candidiasis, HPV, and others) that impair analysis of local adverse effects on the genitalia;
9. Use of topical medications in the genital region that may interfere in the IP evaluation, as well as in its absorption or drug interaction;
10. Possession of penile prosthesis;
11. History of symptomatic hypotension, or diseases that increase the risk of symptomatic hypotension, such as patient with heart diseases (including history of angina and/or heart failure) and nephropathies;
12. Current use of nitrates, such as propatilnitrate (Sustrate®), isosorbide (Monocordil®, Cincordil®, Isordil®), nitroglycerin (Nitradisc®, Nitroderm TTS®, Nitronal®, Tridil®) and isosorbitol dinitrate (Isocord®);ketoconazole; ritonavir; and rifampicin.
13. Findings on ECG and/or laboratory tests that, in the Investigator's criteria, are considered significant and offer risk to the research volunteer's participation or may hinder the study analyses;
14. BP outside the limits considered safe: SBP below 90 mmHg or above 170 mmHg; or DBP below 50 mmHg or above 100 mmHg, except situations such as "white coat syndrome";
15. Diseases that can cause priapism, such as sickle cell anemia, multiple myeloma, or leukemia;
16. Histroy of priapism, defined as painful erection from up to 6 hours.
17. Current relevant diarrhea, defined as duration over four weeks, association with abdominal pain or dysabsortive syndrome, or presence of mucus, pus, or blood in the stool;
18. Known hypersensitivity to tadalafil and/or BZ371A;
19. History of symptomatic Lactose intolorence such as: the necessity of enzymatic treatment, abdominal distension or diarrhea when ingesting products or supplements with lactose;
20. Low adhsesion to 5mg Tadalafil use, characterized by the use of <80% of the pills between the 30th and 60th day post PR;.
21. Pregnant or lacting partner.
22. Partner in childbearing age which does not accept to get exposed to the treatment
23. Any disease, condition or physical finding that the Investigator considers significant and that increases the risk of the research subject's participation or may interfere with the results, including severe debilitating illness, presence of cancer other than prostate cancer, severe mental illness persistent medication abuse;

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Assisted Erectile Function | From up to 30 days before Baseline, Baseline, 30 days, 60 days
  Measurement of the ability to to have an erection that allows sexual intercourse, under use of medication. This will be assessed by using the IIEF questionnaire, domain A (erectile function section) (IIEF-EF).

SECONDARY OUTCOMES:
Change in successful vaginal intercourse rate | From up to 30 days before Baseline, Baseline, 30 days, 60 days
  Rate of successful vaginal intercourse will be assessed through question 3 of the SEP (Sexual Encouter Profile) questionnaire.
Change in quality of sexual intercourse | 30 days, 60 days
  Quality of sexual intercourse, through the EDITS questionnaire (Erectile Dysfunction Inventory of Treatment Satisfaction);
Change in penile extension | Baseline, 30 days, 60 days
  Penile extension, measured with a ruler.
Penile Blood flow increase | From up to 30 days before Baseline, Baseline, 30 days, 60 days
  Increased blood flow, assessed by peak systolic velocity (PSV), end-diastolic velocity (EDV) and resistivity index (RI) assessed by Doppler examination;
Adverse effects report | Baseline 30 days, 60 days and 75 days
  Adverse effects evaluation of compound use and application
Physical examination of the applied region | From up to 30 days before Baseline, Baseline, 30 days, 60 days and 75 days
  Number of participants with abnormal physical exam findings in the applied region
Change in SBP | From up to 30 days before Baseline, Baseline, 30 days, 60 days and 75 days
  Change in Systolic Blood Pressure
Change in DBP | From up to 30 days before Baseline, Baseline, 30 days, 60 days and 75 days
  Change in Diastolic Blood Pressure
Change in Heart Rate (HR) | From up to 30 days before Baseline, Baseline, 30 days, 60 days and 75 days
  Change in Heart Rate
Basal chest electrocardiogram (ECG). | From up to 30 days before Baseline, 30 days and 60 days
  Number of participants with abnormal ECG test results
Blood evaluation | From up to 30 days before Baseline, and 60 days
  Number of participants with abnormal laboratory test results
Urine evaluation | From up to 30 days before Baseline, and 60 days
  Number of participants with abnormal laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Otávio Torres, Dr, Principal Investigator — Hospital Urológica
Locations (1):
- Hospital Urológica, Belo Horizonte, Brazil